CLINICAL TRIAL: NCT05028530
Title: Correlation Analysis of Lens Nucleus Density and Surgical Parameters Based on Long-range Swept-source Optical Coherence Tomography and Scheimpflug Technology
Brief Title: Correlation Analysis of Lens Nucleus Density and Surgical Parameters Based on Ss-oct and Scheimpflug Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: LZL nucleus density
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Age-related Cataract
Keywords: cataract; nucleus density; phacoemulsification parameters; ss-oct; scheimpflug
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the correlation between three different lens nuclear opacity classification methods and intraoperative phacoemulsification parameters .

DETAILED DESCRIPTION:
Slit-lamp lens images, Pentacam and IOL-Master 700 images were collected in patients with dilated pupil before cataract surgery, and phacoemulsification parameters on the Centurion phacoemulsification machine (Alcon) screen were recorded. Spearman correlation analysis was used to analyze the correlation between lens nuclear density and phacoemulsification parameters based on SS-OCT and Scheimpflug techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Age-related cataracts performed by the same surgeon in our hospital;
2. Pupil diameter can be enlarged more than 6 millimetre.

Exclusion Criteria:

1. The pupil diameter cannot be dilated greater than 6mm;
2. previously ocular surgery or laser treatment;
3. history of ocular trauma;
4. other ocular diseases such as keratoconus, glaucoma and retinal detachment;
5. corneal opacities caused by leucoma, pterygium and other diseases;
6. lens dislocation or complicated cataract surgery (any complications during/after the operations);
7. poor fixation leading to low image quality or inability to cooperate with examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study, age-related cataract patients who met the criteria for cataract surgery and underwent cataract surgery by the same surgeon in our hospital were included.
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Lens nuclear opalescence(NO) and nuclear colour (NC) | 2021.12.30
  After the maximumly pupil dilation, the same experienced ophthalmologist examined all the eyes with slit-lamp digital cameras in dark conditions and scored the lens nuclear opalescence(NO) and nuclear colour (NC) on a scale of 0.1-6.9 according to LOCS III criteria.
Pentacam mean nuclear density (PND) | 2021.12.30
  After the maximumly pupil dilation, Pentacam HR was used to acquire the Scheimpflug images of the lens, and the average density reading for the entire nucleus provided by PNS function was defined as Pentacam mean nuclear density (PND), ranging from 0% to 100%.
Mean nucleus density (MND) of the lens presented by IOL-Master 700 | 2021.12.30
  After the maximumly pupil dilation, the inspected eyes are asked to focus on the indicator light to obtain a high-definition image of the lens. The image is derived to the ImageJ software, and the contour of the lens nucleus is manually drawn. The pixel density of the image within the contour is measured, with a value range of 0-255.The mean pixel density within the region was used to represent the mean nucleus density (MND) of the lens presented by IOL-Master 700.For each eye, the SS-OCT nucleus density is defined as the average of six readings from the corresponding image.
Intraoperative phacoemulsification parameters | 2021.12.30
  The intraoperative phacoemulsification parameters on the Centurion phacoemulsification machine (Alcon) screen were recorded after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Wang W, Zhang J, Gu X, Ruan X, Chen X, Tan X, Jin G, Wang L, He M, Congdon N, Liu Z, Luo L, Liu Y. Objective quantification of lens nuclear opacities using swept-source anterior segment optical coherence tomography. Br J Ophthalmol. 2022 Jun;106(6):790-794. doi: 10.1136/bjophthalmol-2020-318334. Epub 2021 Jan 13. PMID 33441322
- [Background] Makhotkina NY, Berendschot TTJM, van den Biggelaar FJHM, Weik ARH, Nuijts RMMA. Comparability of subjective and objective measurements of nuclear density in cataract patients. Acta Ophthalmol. 2018 Jun;96(4):356-363. doi: 10.1111/aos.13694. Epub 2018 Mar 25. PMID 29575599
- [Background] Lim SA, Shin JY, Chung SH. Useful Prediction of Phacodynamics by Scheimpflug Lens Densitometry in Patients over Age 70. Semin Ophthalmol. 2017;32(4):482-487. doi: 10.3109/08820538.2015.1120756. Epub 2016 Apr 19. PMID 27092580
- [Background] Gupta M, Ram J, Jain A, Sukhija J, Chaudhary M. Correlation of nuclear density using the Lens Opacity Classification System III versus Scheimpflug imaging with phacoemulsification parameters. J Cataract Refract Surg. 2013 Dec;39(12):1818-23. doi: 10.1016/j.jcrs.2013.05.052. PMID 24286839
- [Background] Chen D, Li Z, Huang J, Yu L, Liu S, Zhao YE. Lens nuclear opacity quantitation with long-range swept-source optical coherence tomography: correlation to LOCS III and a Scheimpflug imaging-based grading system. Br J Ophthalmol. 2019 Aug;103(8):1048-1053. doi: 10.1136/bjophthalmol-2018-312661. Epub 2018 Oct 12. PMID 30315132
- [Background] Panthier C, de Wazieres A, Rouger H, Moran S, Saad A, Gatinel D. Average lens density quantification with swept-source optical coherence tomography: optimized, automated cataract grading technique. J Cataract Refract Surg. 2019 Dec;45(12):1746-1752. doi: 10.1016/j.jcrs.2019.07.033. PMID 31856985
- [Background] Panthier C, Burgos J, Rouger H, Saad A, Gatinel D. New objective lens density quantification method using swept-source optical coherence tomography technology: Comparison with existing methods. J Cataract Refract Surg. 2017 Dec;43(12):1575-1581. doi: 10.1016/j.jcrs.2017.09.028. PMID 29335103